CLINICAL TRIAL: NCT00462020
Title: Intravenous Versus Intravenous/Oral Antibiotics for Perforated Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07 02 031
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Results first posted 2011-12-13 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Perforated Appendicitis
Keywords: appendicitis, perforation, abscess, treatment
MeSH Terms: conditions — Appendicitis; Abscess | interventions — Anti-Bacterial Agents; Ceftriaxone; Metronidazole; Home Care Services; Ampicillin; Clavulanic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 5 days of IV antibiotics after appendectomy
  Interventions: Drug: 5 days of IV antibiotics (ceftriaxone and metronidazole)
- 2 (Experimental): home on oral antibiotics to complete 7 days of treatment when tolerating PO's
  Interventions: Drug: Home with oral antibiotics when eating (ampicillin/clavulanic acid)

INTERVENTIONS:
Drug: 5 days of IV antibiotics (ceftriaxone and metronidazole) — 5 days of IV antibiotics (ceftriaxone and metronidazole once a day dosing)
  Arms: 1
Drug: Home with oral antibiotics when eating (ampicillin/clavulanic acid) — Augmentin 40mg/kg BID when tolerating POs to complete 7 days total
  Arms: 2

SUMMARY:
The objective of this study is to scientifically evaluate two different management strategies for perforated appendicitis.

The hypothesis is that early discharge with oral antibiotic therapy may result in a dramatic decrease in medical care expenses for the patient.

The primary outcome variable between the two strategies is abscess rate.

DETAILED DESCRIPTION:
This will be a single institution, prospective, randomized clinical trial involving patients who present to the hospital with perforated appendicitis. This will be a definitive study.

Power calculation was based on abscess rate in the previous prospective, randomized study we just finished. Our current rate is 18%, or just under one-fifth of the patients. A doubling of this rate to 36% would place just over one third of the patients at risk which would be unacceptable. Using a delta of 0.18 with alpha of 0.05 and power of 0.8, the sample size is 74 patients in each arm. Therefore we will anticipate enrolling 150.

Subjects will be those children who undergo a laparoscopic appendectomy as part of their routine care.

Perforation will be defined as an identifiable hole in the appendix or stool in the abdomen.

The control group will receive current standard care: ceftriaxone 50mg/kg once a day (maximum dose = 2 grams) and metronidazole 30mg/kg once a day (maximum dose = 1 gram) with once a day dosing for both. The length of antibiotic therapy will be a minimum of 5 days. At that time, if they have been afebrile for at least 24 hours, a white blood cell (WBC) count will be obtained, and if that is within normal limits, the antibiotics will be discontinued and the patient will be discharged. If the WBC is elevated, they will receive another 2 days before recheck, if still elevated, they receive another 3 days and a CT Scan is obtained. If, after 5 days of therapy, the patient remains febrile, therapy will continue until afebrile before a WBC check is performed. This is all our current standard management.

The experimental group will receive the same combination of antibiotics while in the hospital. When the patient is tolerating a regular diet, on oral pain medication and has been afebrile for over 12 hours, they will be discharged on oral antibiotics to complete a course of 7 days. The home antibiotic regimen will be ampicillin/clavulanic acid (Augmentin®). Augmentin® dose will be 40mg/kg twice a day. They will be asked to bring their pill containers with them to clinic where we will quantify medication compliance.

Given the purpose of this study is the comparison of oral antibiotics to intravenous antibiotics, an allergy to one of the above medications will not be considered an exclusion criteria. In such cases the patient will be treated with an alternative that offers the same spectrum of coverage, but will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Identifiable hole in the appendix or stool in the abdomen at the time of appendectomy

Exclusion Criteria:

* Known immune deficiency
* Abscess identified on pre-op imaging
* Another condition affecting surgical decision making or recovery (e.g. hemophilia, severe cardiac or respiratory co-morbidities).

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 2007-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn D St. Peter, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients with perforated appendicitis were recruited for this study.
Groups:
- IV Only: 5 days of IV antibiotics after appendectomy
- IV and Oral Abx: home on oral antibiotics to complete 7 days of treatment
Period: Overall Study
Arm/Group | IV Only | IV and Oral Abx
Started | 52 | 50
Completed | 52 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- IV and Oral Abx: home on oral antibiotics to complete 7 days of treatment when tolerating PO's
- Total: Total of all reporting groups
Arm/Group | IV Only | IV and Oral Abx | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 52 | 50 | 102
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (4.2) | 10.1 (4.6) | 9.9 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 43
  Male | 32 | 27 | 59
Region of Enrollment [Number; unit: participants]
  United States | 52 | 50 | 102

OUTCOME MEASURES:

1. Primary Outcome: Abscess After Appendectomy
Time Frame: 1 month
Measure: Number; unit: number of patients
Arm/Group | IV Only | IV and Oral Abx
Number analyzed (Participants) | 52 | 50
number of patients | 10 | 10

2. Secondary Outcome: Operative Time
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | IV Only | IV and Oral Abx
Number analyzed (Participants) | 52 | 50
Minutes | 41.06 (15.36) | 46.30 (19.42)

3. Secondary Outcome: Time to Regular Diet
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | IV Only | IV and Oral Abx
Number analyzed (Participants) | 52 | 50
Hours | 68.00 (35.06) | 61.42 (32.12)

4. Secondary Outcome: Length of Stay After Operation
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | IV Only | IV and Oral Abx
Number analyzed (Participants) | 52 | 50
Days | 6.06 (2.00) | 4.48 (2.36)

5. Secondary Outcome: Total Healthcare Visits
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | IV Only | IV and Oral Abx
Number analyzed (Participants) | 52 | 50
Visits | 3.1 (1.4) | 3.1 (1.2)

ADVERSE EVENTS:
Time Frame: 1 month
Description: No Adverse Events were recorded
Arm/Group | IV Only | IV and Oral Abx
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/50
Other Adverse Events (participants affected / at risk) | 0/52 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes